CLINICAL TRIAL: NCT00534885
Title: The Phase Ⅳ Clinical Trial to Evaluate the Safety, Immunogenicity, and Immune Persistence of Three Consecutive Lots of an Inactivated Hepatitis A Vaccine in Healthy Children
Brief Title: Safety, Immunogenicity, and Immune Persistence Study of an Inactivated Hepatitis A Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-HA-4006; PRO-HA-4008 (11 Y follow-up) (Other: Sinovac Biotech Co., Ltd)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis A
Keywords: inactivated hepatitis A vaccine; Healive; safety; immunogenicity; immune persistence
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Healive® Lot 1 (Experimental)
  Interventions: Biological: Healive® Lot 1
- 2: Healive® Lot 2 (Experimental)
  Interventions: Biological: Healive® Lot 2
- 3: Healive® Lot 3 (Experimental)
  Interventions: Biological: Healive® Lot 3
- 4: control vaccine (Havrix) (Active Comparator)
  Interventions: Biological: Havrix

INTERVENTIONS:
Biological: Healive® Lot 1 — Inactivated hepatitis A vaccine manufactured by Sinovac Biotech Co., Ltd.; two-dose regimen with 6 months apart
  Arms: 1: Healive® Lot 1
Biological: Healive® Lot 2 — Inactivated hepatitis A vaccine manufactured by Sinovac Biotech Co., Ltd.; two-dose regimen with 6 months apart
  Arms: 2: Healive® Lot 2
Biological: Healive® Lot 3 — Inactivated hepatitis A vaccine manufactured by Sinovac Biotech Co., Ltd.; two-dose regimen with 6 months apart
  Arms: 3: Healive® Lot 3
Biological: Havrix — Inactivated hepatitis A vaccine manufactured by GlaxoSmithKline Biologicals; two-dose regimen with 6 months apart
  Arms: 4: control vaccine (Havrix)

SUMMARY:
A double-blind, randomized and controlled clinical trial was conducted in healthy children aged from 1 to 8 years to evaluate the immunogenicity and safety of three consecutive lots of a preservative-free inactivated hepatitis A vaccine (Healive®).

Participants who completed their primary vaccination were invited to participate in the follow-up phase. Written informed consents were obtained from them. The follow-up study was open-label. These subjects were visited in the next 11 years for blood sampling and assessment of immune persistence induced by vaccination.

DETAILED DESCRIPTION:
The investigated vaccine is an inactivated, adjuvanted and preservative-free hepatitis A vaccine. Each dose contained 250 U HAV antigen in 0.5 milliliter.

Total 400 subjects were enrolled and assigned into four groups, each receiving one of the three lots of Healive® or an established control vaccine at month 0 and 6. Anti-HAV titers were determined at month 1, 6 and 7. Anti-HAV titer over 20 mIU/ml is defined as seroprotection.

After the full immunization schedule, written informed consents were obtained from subjects who would like to participate in the follow-up study. Blood samples of these subjects were collected at month 18, 30, 42, 54, 66, 112,138 after the first injection to evaluate the seroconversion rates (SCRs) and geometric mean concentrations (GMCs) of antibody against hepatitis A virus. Serological results of the follow-up study were then used to explore suitable statistical model for predicting the persistence of hepatitis A vaccine-induced antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Health children from 1 to 10 years
* Not participate in any other trial during the course of the trial
* Informed consent

Exclusion Criteria:

* Any history of allergic reactions or convulsions following vaccination
* Other known or planned vaccination within 1 month prior to the study and during the study period
* Any chronic illness/disease including virus hepatitis, tuberculosis and epilepsy
* Presence of any congenital abnormality, upgrowth obstacle
* Any history/suspicion/presence of neurology and Lunacy
* Any current or foreseeable use of immunosuppressors (i.e. corticosteroids , immunoglobulins) within 1 month prior to the vaccination and during the period of the study
* Contraindication to intramuscularly injection due to thrombocytopenia or other bleeding disorders
* Abnormal ALT
* Positive markers for anti-HAV and HBV（HBsAg）infection
* Presence of fever at the time of vaccination, i.e. body temperature (by mouth) > 37.0 centigrade.

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2006-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Anti-HAV titer | 7 months after the first dose
  To evaluate the immune responses to the inactivated hepatitis A vaccine by detecting the anti-HAV titer using microparticle enzyme immunoassay (MEIA) assay.

SECONDARY OUTCOMES:
Solicited adverse reactions (AE): local reactions and systematic reactions | 72 hours after each injection
  Solicited AEs were recorded until 72 hours after each injection
Unsolicited adverse reactions (AE) | 7 months after the first dose
  Unsolicited AEs were recorded until month 7
Change of anti-HAV titer: geometry mean titer(GMT) and seroconversion rate | baseline (day 0), month 1, 6, 7, 18, 30, 42, 54, 66,112,138 after the first dose
  Blood samples were collected at day 0, month 1, 6, 7, 18, 30, 42, 54, 66,112, 138 after the first dose to assess the change of long-term immune response. Anti-HAV antibodies were assessed by microparticle enzyme immunoassay (MEIA) assay (cut off: 20 mIU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yu Chen, Principal Investigator — Changzhou City Centre for Diseases Control and Prevention
Locations (1):
- Changzhou City Center for Disease Control and Prevention, Changzhou, Jiangsu, China